CLINICAL TRIAL: NCT01447680
Title: Clinical Trial Comparing Two Types of Blood Samples (Plasma and SMARTplasma) for HIV and HCV Antibody Testing
Brief Title: Comparison of Plasma & SMARTplasma for Human Immunodeficiency Virus (HIV) and Hepatitis C Virus (HCV) Antibody Testing
Status: Completed | Type: Observational
Sponsor: G & W Laboratories Inc. (Industry)
Collaborators: Alquest (Industry); SMART Biotech Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: ST-2011-HIV, Version 4
Record Dates: First submitted 2011-09-22; First posted 2011-10-06 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Human Immunodeficiency Virus Infection; Hepatitis C
Keywords: HIV infection; HCV infection; SMARTube; SMARTplasma
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and SMARTplasma (SMARTplasma is plasma sample from whole blood treated with SMARTstim)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Blood samples, low risk population
- Blood samples, high risk population
- Blood samples, known HIV positive

SUMMARY:
The purpose of this study is to compare the results for HIV and/or Hepatitis C Virus antibody testing when using routine plasma versus SMARTplasma from the same blood sample. SMARTplasma is enriched for antibodies via a stimulation step of whole blood in a SMARTube™ (SMARTstim™ in the USA).

DETAILED DESCRIPTION:
Following exposure to HIV and HCV, there is a "window period" where a person is infected with the virus but does not produce antibodies at a high enough level so they can be detected by antibody detection test methods. During this time, the person is capable of unknowingly transmitting the virus to others. SMARTstim (SMARTube)is a blood sample additive which pre-treats blood, stimulating antibody production in vitro so as to bring it to detectable levels using ELISA (or any other antibody test method). Accelerated antibody production allows antibody detection in specimens that would otherwise be below the detectable limit of antibody test kits. Plasma samples from blood pretreated with SMARTstim are referred to as "SMARTplasma".

A total of 1,600 blood samples will be collected and tested using an ELISA for HIV and HCV using FDA-approved test kits. The populations include:

* 1000 samples from low risk individuals (blood donors) from 3 geographical locations
* 500 samples from high risk individuals at risk for HIV from 2 geographical locations
* 100 known HIV seropositives

This is a non-linked study; that is, no subject identifiers will be associated with the collected blood. Subjects will not receive any correspondences and will not receive any test results.

If discordant results occur between the plasma and SMARTplasma samples, those samples will be retested. A Western Blot will be performed on ELISA repeat reactive discordant samples. HCV testing using an FDA-approved assay may also be performed using retained samples.

Simple statistical methods will be performed as necessary to analyze concordance of results between the sample types in the same ELISA assay.

Secondarily, it is expected that within the scope of this study, it will be shown that:

* Using SMARTplasma does not adversely affect diagnostic specificity of the HIV and/or HCV antibody assay used; i.e., no increase in the rate of HIV or HCV false positive results.
* Using SMARTplasma does not adversely affect diagnostic sensitivity of the HIV and/or HCV antibody assay used; i.e., no decrease in the number of true positive samples.
* Samples from persons with early or acute infection may show a positive result when using SMARTplasma, while those from plasma will test negative.
* SMARTplasma samples using heparin or EDTA collection tubes and the correlating SMARTstim are comparable.
* SMARTplasma samples that have been frozen show comparable results to correlating SMARTplasma samples that have been refrigerated.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-64,
* Are not pregnant
* Not have a life-threatening disease
* Not immunosuppressed (HIV therapy allowed)
* Are able to give consent, and (6) who appear healthy.

Exclusion Criteria:

* Do not meet the inclusion criteria
* Are enrolled in an HIV vaccine study,
* Who have previously been enrolled in this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Laboratory Sample from low risk population (i.e., blood donors), high risk population and known positive patients.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Concordance of positive and negative results between normal and treated plasma samples when both are tested with the same HIV and/or HCV Enzyme Linked Immunosorbant Assay (ELISA) | Blood samples for HIV and HCV testing will be collected at time of consent (day 1).
  There is one timepoint (day 1)for which the primary outcome measure will be assessed and data will be presented. Samples will be collected, delinked and shipped to core lab within 1 day of collection where samples will be processed and subsequently analyzed for HIV and HCV antibodies. Samples will be frozen and retained for future testing. Results of all testing of correlating SMARTplasma and normal plasma samples will be reported as either positive or negative and these results will be compared for concordance.

SECONDARY OUTCOMES:
Sensitivity and specificity of HIV and HCV antibody assays when used with SMARTplasma | Blood samples for HIV and HCV testing will be collected at time of consent (day 1).
  Testing to demonstrate that SMARTplasma does not adversely affect diagnostic specificity & sensitivity of the HIV or HCV antibody assay used (no increase in rate of false positives or false negatives); however,samples from persons with early or acute infection may show a positive result when tested with SMARTplasma while those from normal plasma will test negative. Results of all testing of correlating SMARTplasma and plasma samples will be reported as either positive or negative and these results will be compared for concordance.
Correlation of results from two different sample types (heparin vs EDTA) | Blood samples for HIV and HCV testing will be collected at time of consent (day 1).
  Testing will determine if SMARTplasma samples from collections in heparin or ethylenediaminetetraacetic acid (EDTA) tubes and the correlating SMARTstim sample results are comparable. Results of all testing of correlating heparin and EDTA samples will be reported as either positive or negative and these results will be compared for concordance.
Correlation of results from refrigerated versus frozen then thawed samples | Blood samples for HIV and HCV testing will be collected at time of consent (day 1).
  Following testing for HIV and HCV antibodies (primary outcome measure), an aliquot of each SMARTplasma test samples will be frozen, thawed and retested for HIV and HCV antibodies side-by-side with a corresponding fresh/refrigerated (non-frozen and thawed) sample. Testing will determine if SMARTplasma samples that have been frozen and thawed prior to testing show comparable results to correlating SMARTplasma samples that have been refrigerated. Results will be reported as either positive or negative and these results will be compared for concordance.

CONTACTS AND LOCATIONS:
Overall Officials: Niel Constantine, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (7):
- United States (7):
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - American Red Cross, Douglasville, Georgia
  - Evelyn Jordan Center, Baltimore, Maryland
  - University of Maryland, School of Medicine, Baltimore, Maryland
  - Man Alive, Inc., Baltimore, Maryland
  - Reach (Ibr), Baltimore, Maryland
  - Bellevue Hospital, New York, New York

REFERENCES:
- [Background] Mumo J, Vansover A, Jehuda-Cohen T. Detecting seronegative-early HIV infections among adult versus student Kenyan blood donors, by using Stimmunology. Exp Biol Med (Maywood). 2009 Aug;234(8):931-9. doi: 10.3181/0812-RM-372. Epub 2009 Jun 2. PMID 19491368
- [Background] Pilcher CD, Tien HC, Eron JJ Jr, Vernazza PL, Leu SY, Stewart PW, Goh LE, Cohen MS; Quest Study; Duke-UNC-Emory Acute HIV Consortium. Brief but efficient: acute HIV infection and the sexual transmission of HIV. J Infect Dis. 2004 May 15;189(10):1785-92. doi: 10.1086/386333. Epub 2004 Apr 28. PMID 15122514
- [Background] Novikov I, Jehuda-Cohen T. HIV type 1 infection among Ethiopian immigrants to Israel: enhanced in vitro antibody stimulation for estimating the length of the window period. AIDS Res Hum Retroviruses. 2009 Feb;25(2):165-74. doi: 10.1089/aid.2008.0151. PMID 19239355